CLINICAL TRIAL: NCT03427710
Title: A Placebo-controlled, Single Blind, Randomised, Phase I, First In Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered CiVi007 in Subjects With an Elevated LDL C Level
Brief Title: A First In Human Study to Assess CiVi007 in Subjects With an Elevated LDL-Cholesterol Level
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Civi Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CiVi-001
Record Dates: First submitted 2018-01-31; First posted 2018-02-09 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Adaptive design allowing modifications in single and multidose arms
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort A1 (Experimental): CiVi007 dose 1
  Interventions: Drug: CiVi007
- Cohort A2 (Experimental): CiVi007 dose 2
  Interventions: Drug: CiVi007
- Cohort A3 (Experimental): CiVi007 dose 3
  Interventions: Drug: CiVi007
- Cohort A4 (Experimental): CiVi007 dose 4
  Interventions: Drug: CiVi007
- Cohort A5 (Experimental): CiVi007 dose 5
  Interventions: Drug: CiVi007
- Combined placebo group (Placebo Comparator): group response from placebo subsets of dosing cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CiVi007 — cholesterol lowering drug
  Arms: Cohort A1; Cohort A2; Cohort A3; Cohort A4; Cohort A5
Other: Placebo — matching placebo to CiVi007
  Arms: Combined placebo group

SUMMARY:
The primary objective of the study is to assess pharmacokinetics, dynamics, safety and tolerability of CiVi007 following single and multiple subcutaneous doses in subjects, including those on statin therapy

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, of any race, with fasting LDL C >2.6 mmol/L (100 mg/dL) and fasting serum triglycerides <4.52 mmol/L (400 mg/dL)
* haematology and clinical chemistry without clinically significant abnormal values
* Normal renal and hepatic function
* Women must not be pregnant, lactating or of child bearing potential
* Men must be willing to use appropriate contraception during the study
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Key Exclusion Criteria:

* Any uncontrolled or serious disease, or any medical or surgical condition
* History or presence of coronary heart disease, peripheral artery disease, or cerebrovascular disease
* Uncontrolled hypertension
* Insulin dependent diabetes mellitus
* Secondary dyslipidemia
* History of renal or hepatic diseases, acquired immune deficiency syndrome, positive human immunodeficiency virus test and/or history of viral hepatitis B or C
* History of cancer within 5 years
* History of high alcohol consumption or positive alcohol breath test or urinary test for drugs of abuse
* Participation in another clinical study within 3 months prior to screening or participation in another study
* Use of treatment (e.g. antibody) towards PCSK9
* History of multiple drug allergies or intolerance to subcutaneous injection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
LDL Cholesterol | Maximum post dose within 8 weeks
  % LDL-C reduction

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of CiVi007 | 8 weeks
  Pharmacokinetic Outcome Measure
PCSK9 level | Maximum post dose within 8 weeks
  maximal % reduction in the level of circulating PCSK9

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, Principal Investigator — Covance
Locations (1):
- Leeds Clinic, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided